CLINICAL TRIAL: NCT05585866
Title: Propofol and Sevoflurane Anesthesia in Colorectal Cancer Surgery: Incidence of Acute Kidney Injury
Acronym: PROSACC
Status: Active, not recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: PROSACC2021
Record Dates: First submitted 2022-10-13; First posted 2022-10-19 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Acute Kidney Injury; Cancer Colorectal
Keywords: sevoflurane; propofol; plasma creatinine
MeSH Terms: conditions — Acute Kidney Injury; Colonic Neoplasms | interventions — Anesthetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Sevoflurane: The group of patients which received sevoflurane as randomized anesthetic modality.
  Interventions: Drug: Anesthesia Agent
- Propofol: The group of patients which received propofol as randomized anesthetic modality.
  Interventions: Drug: Anesthesia Agent

INTERVENTIONS:
Drug: Anesthesia Agent — The two anesthetic modalities included intravenous propofol anesthesia and sevoflurane gas anesthesia administered according to standard clinical praxis.

SUMMARY:
The goal of this observational study is to compare anesthetic modalities (intravenous propofol anesthesia with sevoflurane gas anesthesia) in patients who underwent colorectal cancer resection surgery regarding the outcome of acute kidney injury.

The main questions it aims to answer are:

* is there a difference in acute kidney injury incidence in the two anesthetic modalities?
* is there a difference in plasma creatinine between the two anesthetic modalities?
* are there any patient characteristics or intraoperative factors that effect the incidence of acute kidney injury in either anesthetic modality?

The study will analyze data from the CAN clinical trial database. (Cancer and Anesthesia: Survival After Radical Surgery - a Comparison Between Propofol or Sevoflurane Anesthesia, NCT01975064)

ELIGIBILITY:
Inclusion Criteria:

* colorectal surgery and participant in the CAN trial

Exclusion Criteria:

* missing blood samples

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent colorectal cancer resection surgery and gave consent to participate in the CAN trial.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute Kidney Injury | Within 10 days of surgery
  Compare the incidence of AKI (n, %) in the two anesthetic modalities. Number of participants (n, %) with AKI and number of participants (n, %) with AKI stage 1-3 within the different anesthetic modalities at 0-3 days and 4-10 days postoperatively. KDIGO (Kidney Disease: Improving Global Outcome) criteria for plasma creatinine are used as criteria for AKI. The highest value of plasma creatinine within the time frame will be used to define AKI stage.
Changes in plasma creatinine | Within 30 days of surgery
  Changes in plasma creatinine over time in both groups of anesthesia. Plasma creatinine from preoperative, postoperative after 0-3 days, postoperative 4-10 days and after 30 days. Maximum plasma creatinine for each participant at these time point will be used in the regression analysis.

SECONDARY OUTCOMES:
AKI incidence in the cardiovascular disease population | Within 10 days of surgery
  Compare the incidence of AKI (n, %) during the two anesthetic modalities in the population with present cardiovascular disease. Classified according to KDIGO AKI stage 1-3 changes in plasma creatinine. The highest value of plasma creatinine within the time frame will be used to define AKI stage.
Association of sex on AKI incidence | Within 10 days of surgery
  Compare the incidence of AKI (n, %) in men vs women. This analysis will be done in both groups separately and in the entire population independent of anesthetic modality.
Association of age on AKI incidence | Within 10 days of surgery
  Compare the incidence of AKI (n, %) in participants older vs younger than 65. This analysis will be done in both groups separately and in the entire population independent of anesthetic modality.

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No